CLINICAL TRIAL: NCT03732144
Title: Connect Through PLAY: A Staff-based Physical Activity Intervention for Middle School Youth
Acronym: Connect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Nicole Zarrett, Professor of Psychology, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00073309; 1R01NR017619-01 (NIH)
Record Dates: First submitted 2018-10-06; First posted 2018-11-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity; Obesity Prevention
Keywords: Physical Activity; Community-based Intervention; Social Motivational Theories; Behavioral Change; Agents of Change; Social Mechanisms
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The prospective randomized controlled trial is a nested cohort design that compares two levels of the intervention, a staff-based social development PA program to a generalized ASP health curriculum control, over a 10-month (40 week) time period (16-week intervention, 6 month followup). A total of 30 ASPs serving underserved middle school (~40 youth and ~5 staff per school; N=1200 youth, 150 staff) will be randomly assigned to either receive the Connect intervention or serve as the standard ASP Health curriculum control. The project will be implemented over a 5-year period with a new cohort of 6 ASPs added each year (a total of 5 cohorts, with 6 ASPs in each cohort).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect Staff-based PA intervention (Experimental): Sites receiving the Connect physical activity intervention will involve three related components - a staff health promotion initiative that helps staff pursue personally-tailored health goals and involves weekly 'check-ins', a tailored social PA curriculum to implement within the program's enrichment hour at least 3 times per week, and a comprehensive staff training program that provides strategies and tools for improving social connections within the program and guided support for implementing the social PA curriculum.
  Interventions: Behavioral: Connect Staff-based PA intervention
- Connect Health Curriculum Control (Other): Sites receiving the general health curriculum control will also involve three related components- a comprehensive health program curriculum that includes activities that are interactive and fun and where students will learn about a variety of health behaviors (nutrition, stress reduction, etc.) and life skills through group activities, a staff training program that provides strategies and tools for implementing program curriculum, and on-going support from the Connect staff.
  Interventions: Other: Connect Health Curriculum Control

INTERVENTIONS:
Behavioral: Connect Staff-based PA intervention — After school program sites receiving the Connect intervention will receive a 16 week program that includes three related components - a staff health promotion initiative that helps staff pursue personally-tailored health goals and involves weekly 'check-ins', a tailored social PA curriculum to implement within the program's enrichment hour at least 3 times per week, and a comprehensive staff training program that provides strategies and tools for improving social connections within the program and guided support for implementing the social PA curriculum. Compared to control ASPs, ASPs receiving the 'Connect' program are expected to show greater improvements from baseline to post- and 6 mo follow-up in PA-related social mechanisms, youth PA, and staff PA.
  Other Names: Connect through PLAY
  Arms: Connect Staff-based PA intervention
Other: Connect Health Curriculum Control — After school program sites receiving the general ASP health curriculum control will address the prevention of several negative health behaviors (e.g., substance use, stress, etc) and also involve three related components- a comprehensive health program curriculum that includes activities that are interactive and fun and where students will learn about a variety of health behaviors (nutrition, stress reduction, etc.) and life skills through group activities, a staff training program that provides strategies and tools for implementing program curriculum, and on-going support from the Connect staff. This arm will serve as the comparison group to the Connect Staff-based PA intervention
  Other Names: Connect through PLAY
  Arms: Connect Health Curriculum Control

SUMMARY:
The overall goal of the Connect Through Positive Leisure Activities for Youth (PLAY) Project is to improve staff capacity for implementing effective physical activity (PA) programming within middle school after school programs serving high-risk youth. All components of the 'Connect' intervention (health promotion initiative, comprehensive training, and tailored physical activity curriculum) aim to support staff cohesion, motivation and efficacy in facilitating a PA context that supports youth social goals and meaningful connections. To this end, the investigators will be implementing a 5-year randomized controlled trial with 30 ASPs. Compared to control programs, after school programs receiving the 'Connect' program are expected to show greater improvements from baseline to post- and 6 mo follow-up in social mechanisms, youth PA, and staff PA. The Connect through PLAY project will provide important insights into what supports are needed (and efficacious) for after school program staff to create a positive social climate to promote increases in youth motivation and participation in physical activity.

DETAILED DESCRIPTION:
Although after school programs (ASPs) have been recognized as a critical context for promoting youth physical activity (PA), with broad reach to underserved communities, research by the Principal Investigator and others have indicated that ASPs continue to struggle to meet policy guidelines for daily youth PA. Moreover, despite continued increases in obesity rates among U.S. adolescents, there have been few ASP interventions focused on underserved adolescents, and limited-to-no impact on adolescents' sustained behavior change. Previous ASP studies by the PI demonstrate that social mechanisms overlooked in previous interventions (e.g., developing friendship and connection to peers and staff through PA; group belonging, including positive peer PA norms and tangible support) are key predictors of youth PA. The research team recently completed a feasibility trial (NIH R21 HD077357) within 6 ASPs (3 intervention vs. 3 standard- health curriculum controls) for underserved middle school youth that was the first intervention to date to address these youth PA social goals/mechanisms. Findings showed positive effects for changing staff behaviors, improving youth PA social supports and connections with peers and staff, and increasing youth PA. The proposed study will expand on the previous ASP feasibility trial with a novel translational approach that works with pre-existing ASPs and targets staff as instrumental for sustainable changes in social mechanisms within the ASP setting for increasing the daily PA of underserved adolescents. The proposed project will be a prospective, randomized controlled trial comparing a staff-based social development PA program to a standard ASP health curriculum control. The proposed efficacy trial will enhance the influence of pre-existing ASP staff as key change agents and address social developmental needs of adolescents overlooked in previous interventions through employing a novel theoretical framework that expands on social developmental theory and the social mechanisms highlighted by Self-Determination Theory, Achievement Goal Theory, and Social Cognitive Theory. The intervention will target the three key social mechanisms of "PA social affiliation goals" for increased and sustained PA of staff and underserved middle school youth (i.e., Friendships/connections through PA; Group Belonging, and; Staff Connection). All components of the intervention (health promotion initiative, comprehensive training, and tailored social PA curriculum) aim to improve staff capacity for facilitating a PA context that supports these social goals/mechanisms (connections, group belonging) and increases the influence of ASP staff as positive PA role models and agents of change.

Compared to control ASPs, ASPs receiving the 'Connect' program are expected to show greater improvements from baseline to post- and 6 mo follow-up in social mechanisms, youth PA, and staff PA. The results of this proposed project will demonstrate the efficacy of the intervention, and will assist in developing a model of training, motivating, and empowering ASP staff to address social mechanisms that promote youth PA for conducting a large scale effectiveness trial.

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* Must be currently enrolled in the after school program
* Have parental consent to participate
* Agree to study participation (assent)
* Be available for baseline and post-intervention measurement.

Inclusion for Adults (Program Staff):

* Must be part of the after school staff
* No medical condition or disorder that would limit participation
* Available and able to participate in the data collection and the intervention phase (trainings, health initiative, etc) for the study period.

Exclusion Criteria for Adolescents and Adults (Program Staff)

* Have a medical condition that would interfere with the prescribed physical activity intervention plan
* Have a developmental delay or are in treatment for a psychiatric disorder such that the intervention materials will not be appropriate.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1350 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Greater increases (change) in physical activity (i.e., light, moderate, vigorous PA; using 7-day omni-directional accelerometers) of youth and staff receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6mo follow-up
  Objective assessments of PA will be obtained on both staff and youth with omni- directional accelerometers. Data will be recorded in 30-s epochs to best capture short bouts of vigorous activity and raw activity data will be converted into time spent in light PA (1.6-2.9 metabolic equivalents (METS); count cut points=100 and 1500 for youth and 110-1534 for adults) and moderate-to-vigorous (MV)PA (3-8.9 METS; counts ≥ 1500 for youth and ≥ 1535 for adults) based on activity count thresholds for youth (identified by Puyau et al.) and adults (identified by Wilson, Co-I and Troiano et al) respectively. Youth and staff will wear the belts for one full week at baseline, the 8 wk intervention midpoint, 16 week endpoint, and 6 mo follow-up.

SECONDARY OUTCOMES:
Greater improvements (change) in the Connect Staff-based PA intervention ASPs compared to General Health Curriculum control in targeted social mechanisms within the ASP for promoting physical activity using a social climate observation tool | baseline to 6mo follow-up
  Systematic observations will be conducted using the System for Observing Children's Activity and Relationships during Play (SOCARP) and a supplemental social climate observation tool that has been developed and tested by the PI (MCOT-PA). Key social mechanisms assessed include youth peer interactions and social behaviors (e.g., prosocial interactions like praising peers, antisocial interactions like teasing/bullying), staff behaviors and interactions with youth (e.g., providing praise; engaging in PA with youth), and the nature of activities for supporting connection and belongingness (e.g., inclusive). Consistent with other PA interventions, teams of two coders will make continuous observations of daily activities throughout 5 days at each ASP at baseline, 8wk midpoint, 16wk endpoint, and 6mo follow-up.
Greater improvements (change) in targeted youth PA-based social motivational outcomes of youth receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6mo follow-up
  Changes in social, cognitive, and affective components of youth PA motivations will be assessed. Improvements in PA social motivations will be measured using The Social Motivational Orientations Scale for Sport (SMOSS) which assesses youth's social affiliation orientation toward PA (7 items; 5pt scale: 1=strongly disagree, 5=strongly agree; M=2.44; SD=1.04; reliability coefficients range from .77 to .87), with higher mean scores on the affiliation sub scale indicating greater affiliation goals for PA participation.
Greater improvements (change) in targeted youth PA-based cognitive motivational outcomes of youth receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6mo follow-up
  Changes in social, cognitive, and affective components of youth PA motivations will be assessed. Youth cognitive components of PA motivation will be assessed using the Treatment Self-Regulation Questionnaire (15 items; 7pt scale: 1=not at all true for me [not autonomously regulated], 7=very true for me; reliability coefficient= .73) autonomous motivation/regulation for exercise, with higher mean scores across scale items indicating greater autonomous regulation.
Greater improvements (change) in targeted youth PA-based affective motivational outcomes of youth receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6mo follow-up
  Changes in social, cognitive, and affective components of youth PA motivations will be assessed. The Affective component of motivation will be assessed using The Intrinsic Interest and Regulatory Motives Scale (reliability coefficients from .83 to .94; 5-pt scale: 1=very false [does not enjoy], 5= very true; M=3.7, SD=1.0) with higher mean scores across scale items indicating youth greater intrinsic enjoyment and degree of affective engagement in exercise.
Greater improvements (change) in youth-staff PA-based social connections for promoting physical activity among youth receiving the Connect Staff-based PA intervention compared to youth in the General Health Curriculum control. | baseline to 6mo follow-up
  Changes in youth PA-based social connections will be measured at three levels: youth-staff connections, peer social connections, and peer support for PA. The Perceived teacher support scale (reliability coefficient =.84; 5-pt scale: 1=completely false [not supportive relationship], 5=completely true [very supportive relationship]; M=3.22; SD=1.05) will be used to evaluate improvements in staff-youth connections, with higher mean scores across the scale items indicating higher quality staff-youth connections.
Greater improvements (change) in youth PA-based peer social support among youth receiving the Connect Staff-based PA intervention compared to youth in the General Health Curriculum control. | baseline to 6mo follow-up
  The Social Support and Exercise Survey (reliability coefficients= .80-.87; short form, 4 items; 5pt scale: 1=never [receive support], 5=very often [receive support]) will be used to measure increases in youth PA-based peer social support, with higher mean scores indicating greater peer support for PA.
Greater improvements (change) in youth PA-based positive peer connections among youth receiving the Connect Staff-based PA intervention compared to youth in the General Health Curriculum control. | baseline to 6mo follow-up
  The Need for Relatedness Scale (reliability coefficients=.86-.92; 7-pt scale: 1-strongly disagree, 5=strongly agree:, M=3.74; SD=.75) will be used to assess youth's own personal experiences with positive peer connections within the program, with higher mean scores across scale items indicating greater positive peer connections.
Document the Fidelity of the Connect program through changes in Staff's collective capacity to lead youth in PA activities within ASPs receiving the Connect Staff-based PA intervention. | baseline to 6 mo follow-up
  Changes in Staff's collective capacity to lead youth in PA activities will be measured through structured interviews using a Readiness Assessment Tool that the PI has developed and tested which examines motivation for implementing the Connect intervention, innovation-specific capacity for Connect (e.g., staff efficacy), and general capacity (e.g., staff cohesion, support and positive relations with higher administration, and overall work satisfaction). The assessment will be conducted at baseline to identify and address any initial program barriers that would impede adoption of the intervention, and again at 8wks (midpoint), 16 wks (endpoint), and 6mo follow-up to determine whether any modifications to implementation are needed to improve adoptability post-intervention.
Greater improvements (change) in targeted staff PA motivational outcomes of staff receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6 mo follow-up
  Staff PA motivation and value will be measured using the Behavioral Regulation in Exercise Questionnaire (BREQ; subscale reliability coefficients range from .78-.90; 24 items; 5pt scale; 0=not true; 4=very true for me), with higher mean scores across scale items indicating greater PA motivation. The assessment will be conducted at baseline, 8wks (midpoint), 16 wks (endpoint), and 6mo follow-up.
Greater improvements (change) in targeted staff PA self-concept and efficacy to overcome barriers of staff receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6 mo follow-up
  Staff PA self-concept and efficacy to overcome barriers impeding their accrual of daily recommended amounts of PA will be measured using the Self Concept and Motivation to Exercise Scale (reliability coefficients range from .63-.90; 7 items; 6pt scale; 0=strongly disagree; 6=strongly agree), and the Self-Efficacy for Exercise Questionnaire (reliability coefficient = .96; 10 items; 5pt scale; 1-not at all confident; 5=extremely confident), respectively. Higher mean scores across the scale items will indicate greater PA self-concept/efficacy. The assessment will be conducted at baseline, 8wks (midpoint), 16 wks (endpoint), and 6mo follow-up.
Greater improvements (change) in staff PA-based social support among staff receiving the Connect Staff-based PA intervention compared to General Health Curriculum control. | baseline to 6 mo follow-up
  The Social Support and Exercise Survey (reliability coefficient .80-.87; 20 items; 5pt scale; 0=none; 4=very often) will assess changes in staff connectedness/support to be active, with higher mean scores across items indicating greater social support. The assessment will be conducted at baseline, 8wks (midpoint), 16 wks (endpoint), and 6mo follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Zarrett, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Deng A, Zarrett N. Examining variations in perceived barriers and self-efficacy for physical activity among adults in underserved communities. J Behav Med. 2026 Jan 19. doi: 10.1007/s10865-025-00627-1. Online ahead of print. PMID 41553615
- [Derived] Deng A, Zarrett N, Sweeney AM. The mediating effects of motivation on the relations between occupational stress and physical activity among underresourced afterschool program staff. BMC Public Health. 2024 Jan 30;24(1):327. doi: 10.1186/s12889-024-17800-x. PMID 38291408
- [Derived] Deng A, Zarrett N, Moon J, Sweeney AM. Changing trajectory of daily physical activity levels among at-risk adolescents: influences of motivational mechanisms. BMC Public Health. 2023 Oct 25;23(1):2089. doi: 10.1186/s12889-023-16949-1. PMID 37880639